CLINICAL TRIAL: NCT04051060
Title: Evaluation of Exercise Capacity and Activity Role Adequacy in Patients With Adult Bronchial Asthma
Acronym: ASTHMA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HÜSNA GÜZEL, Principal İnvestigator, Hacettepe University
Other Study IDs: GO 19/37
Record Dates: First submitted 2019-04-21; First posted 2019-08-09 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Asthma; Activity Role Qualification; Fear of Movement
MeSH Terms: conditions — Asthma; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Bronchial Asthma
- Healthy individuals

SUMMARY:
The aim of this study was to evaluate exercise capacity and activity role adequacy in patients with adult bronchial asthma.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease characterized by increased airway sensitivity to various stimuli and reversible airway obstruction. Asthma is a disease with high morbidity and mortality despite all advances in pathogenesis, diagnosis and treatment in the world. It is estimated that there are approximately 300 million asthmatic patients in the world. In our country, approximately one out of every 12-13 adults and one in 7-8 children have asthma. Clinical symptoms of asthma include shortness of breath, wheezing, coughing. Increased symptoms in asthmatic patients lead to impaired respiratory function. In chronic respiratory problems, participants restrict their activity to avoid shortness of breath. As a result, physical fitness levels are reduced, shortness of breath occurs at earlier workloads, and participants do less activity. In chronic disorders, managing the disease alone may not be enough to optimize normal functioning in daily life. In literature, it is seen that daily life activities, quality of life, school performance and work performance are affected in asthmatic patients. it is thought to be useful in determining the course of treatment to be given to the patient in the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with bronchial asthma by a chest physician
* Being between the ages of 18-65
* Being in a stable period
* Work in the last 12 months

Exclusion Criteria:

* Severe chronic disease other than bronchial asthma (cancer, chronic obstructive pulmonary disease, chronic heart failure, neurological disease, etc.).
* Any physical disability that prevents walking
* Unable to comply with tests
* lack of reading, speaking and writing in Turkish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who will participate in the study will have stable bronchial asthma who is diagnosed in Kocaeli University Faculty of Medicine, Department of Chest Diseases or has a clinical condition that comes to routine control of Cardiopulmonary Rehabilitation Unit of Hacettepe University Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Exercise Capacity | Day 1
  Exercise capacity will be evaluated with a six-minute walk test (6MWT). The patients will be asked to walk as fast as they can in their own walking tempo for six minutes in a 28-meter straight corridor.6DYT distance value has normal values according to age and sex.
  These values will be taken as reference in the interpretation of the measurements.
Evaluation of Activity-Role Adequacy | Day 1
  Activity-role adequacy in asthma patients will be assessed using the "Activity Self-Assessment" questionnaire. The Activity Self-Assessment questionnaire is a person-centered assessment tool designed to determine how illness and disability affect individuals' activities and roles. The Activity Self-Assessment Questionnaire is a person-centered assessment questionnaire consisting of 21 items and importance related to activity-role competence. The Activity Self-Assessment questionnaire asks the individual to score each item and value on two separate 4-point scales for activity adequacy. The points obtained are summed up to obtain two separate total points, namely competence and importance. These scores are converted to scores between 0-100 with the method in the application guide of the scale. As the total score increases, activity self-efficacy and importance increases.

SECONDARY OUTCOMES:
Assessment of Respiratory Functions | Day 1
  Pulmonary function test results will be obtained from hospital records. Pulmonary function test parameters will be expressed as a percentage of expected values by age, height, body weight and gender.
Evaluation of Functional Capacity | Day 1
  The functional capacity of the cases will be evaluated by 30-second sit-up test.The full number of starts is recorded for 30 seconds.
Evaluation of Daily Living Activities | Day 1
  Daily living activities of the patients will be evaluated with the London Chest Daily Living Activities Scale. It is a simple and standardized questionnaire developed for the evaluation of dyspnea caused by activities of daily living in patients with obstructive pulmonary diseases (30). This questionnaire consisting of 15 items; personal care (4 items-dry, dress up upper body, wear shoes / socks, wash hair), housework (make 6 item-bed, change bed linen, window / curtain wash, clean / remove dust, wash dishes, sweep), physical activity (2 items-stair climbing, leaning) and leisure (3 items-walking in the house, socially go out, talk) consists of four components. Each item is given a score ranging from 0 to 5. Higher scores indicate that the limitation in GYA is higher. Scale; total score, component score and question score. The total score can reach up to 75.
Evaluation of Quality of Life | Day 1
  Health-related quality of life will be determined by the Nottingham Health Profile (NHP). The NHP consists of 38 items which one can self-complete without the need for an interviewer. The questionnaire has six subscales: energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items) and physical mobility (8 items). For each subsection there is a possible range of points ranging from 0-100 points. Higher scores indicate more limitations in quality of life.
Assessment of Quality of Life in Asthmatic Patients | Day 1
  The Asthma Specific Quality of Life Questionnaire (AQLQ) developed by Juniper et al. The questionnaire consists of 32 questions, 11 of which are activity restriction, 12 are symptoms, 5 are mood and 4 are environmental exposure. Patients are asked to remember their experience during the previous 2 weeks and to score each item on a 7-point scale. The overall AQLQ score is the average response to 32 questions. In this survey, which is grouped under four main headings, firstly the average score is calculated for each title and then the average of these 4 is considered as the overall quality of life score.
Evaluation of fear of motion | 1st Day
  Kinesiophobia will be determined using the Tampa Kinesiophobia Scale. The Tampa Kinesiophobia Scale is a checklist of 17 questions. The scale uses a 4-point Likert score (1 = Strongly disagree, 4 = Strongly agree). The person gets a total score between 17-68. The higher the score of the person on the scale, the higher the kinesiophobia.
Psychosocial Assessment | Day 1
  Psychosocial status of asthmatic patients will be evaluated using Hospital Anxiety and Depression (HAD) Scale. The survey's validity and reliability study in Turkey Aydemir et al. (1997). This scale is used for diagnosing anxiety and depression in a short time and for determining the risk group, not for diagnosing patients with physical illnesses and those applying to primary health care services. The scale consists of a total of 14 items and the items are 4-point Likert type. HAD-A evaluates anxiety with 7 questions and HAD-D evaluates depression with 7 questions. The lowest score that the patients could get from both subscales was 0 and the highest score was 21. The cut-off points of the HADS Scale were 10 for the anxiety subscale (HAD-A) and 7 for the depression subscale.

CONTACTS AND LOCATIONS:
Overall Officials: MELDA SAĞLAM, PhD, Study Director — Hacettepe University
Locations (1):
- Melda Sağlam, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes